CLINICAL TRIAL: NCT02163629
Title: Impact of Stress Management Training on Quality of Life and Cardiac Post-transplantation Complications in a Controlled Multicentric Comparative Study.
Brief Title: Impact of Stress Management Training After Cardiac Transplantation
Acronym: QUIET
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-842
Record Dates: First submitted 2014-05-27; First posted 2014-06-13 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Heart Transplant
Keywords: Psychotherapeutic intervention; stress management; cardiac transplantation; quality of life

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- psychotherapeutic intervention (Experimental): The psychotherapeutic intervention "stress management" is based on therapeutic, behavioral and cognitive strategies. They are active and put the patient "actor" of his "adaptation" of the heart transplantation entire process. The approached components are emotional, cognitive and behavioral (techniques of communication and problem solving).
  Interventions: Behavioral: Stress management
- Usual medical care (No Intervention)

INTERVENTIONS:
Behavioral: Stress management
  Other Names: The program of "stress management" will include six group sessions at a rate of one session of 2 hours every 15 days. 6 components will be approached:; - stress and relaxation; - cognitive strategies of the stress adaptation; - communication techniques and stress; - problem solving techniques and stress; - stress adaptation; - generalization of stress management in everyday situations
  Arms: psychotherapeutic intervention

SUMMARY:
In spite of major medical advances in heart transplant patients, psychiatric comorbidity remains very high in pre-and post-transplant phases. Anxiety and depression are especially frequent. They impact significantly morbidity and mortality. Especially because they are associated with poor therapeutic adherence and risks of infection and rejection. The inability to make beneficial therapeutic choice can be explained by the negative perception of events, associated with anxio-depressive disorders. This results in an important deterioration in quality of life of patients.

The investigators assume that better management of emotions might reduce the stress of waiting situation and its psychopathological and somatic consequences pre-and post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Men and women on the cardiac transplantation waiting list
* Patients aged 18 years and older
* Signed written informed consent
* Patients under the social security
* Patients with a somatic condition allowing travels
* Patients mastering the French language
* Class II or III NYHA patients

Exclusion Criteria:

* Patients minor or under protection measures
* Patient who have not signed written informed consent
* Patients not mastering the French language
* Patients with psychiatric illness characterized by the axis 1 of DSM IV R
* Patients receiving a psychotherapy or with a psychiatric care
* class IV NYHA patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of a psychotherapeutic intervention on the quality of life of cardiac transplant patients. | The quality of life is evaluated before the cardiac transplantation and during the 12 months after the cardiac transplantation.
  The quality of life is assessed with the MLHFQ - Minnesota Living with Heart Failure Questionnaire.

SECONDARY OUTCOMES:
Anxiety manifestations pre-and post-transplant | Before the cardiac transplantation and during 12 months after the cardiac transplantation
  Anxiety manifestations pre-and post-transplant measured with the State-Trait Anxiety Inventory
Depressive symptoms pre-and post-transplant | Before the cardiac transplantation and during 12 months after the cardiac transplantation
  depressive symptoms pre-and post-transplant measured using the Beck Depression Inventory (BDI-II)
Pre and post-transplant major clinical events | Before the cardiac transplantation and during 12 months after the cardiac transplantation
Hospitalization modalities around the graft | Before the cardiac transplantation and during 12 months after the cardiac transplantation
  by measuring the duration of stay in hospital, number of surgery necessary
Somatic complications after the heart transplantation | During 12 months after the cardiac transplantation
  by measuring the mortality rate and number of graft rejection
The therapeutic adherence pre-and post-transplant | Before the cardiac transplantation and during 12 months after the cardiac transplantation
  using an adherence questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed SAOUD, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Service de Psychiatrie d'Adultes Liaison/Consultation,, Bron
  - Pôle de Psychiatrie et de Neurologie, Grenoble